CLINICAL TRIAL: NCT04477668
Title: Helmet Non-Invasive Ventilation for COVID-19 Patients
Acronym: Helmet-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: King Abdulaziz Medical City, Riyadh, Saudi Arabia (Unknown); King Fahd Hospital of the University, Al Khobar, Saudi Arabia (Unknown); Aseer Central Hospital, Abha, Saudi Arabia (Unknown); King Faisal Specialist Hospital & Research Center (Other); King Fahad Hospital, Madinah, Saudi Arabia (Unknown); Al Amiri Hospital, Kuwait (Unknown); King Abdulaziz University (Other); King Saud Medical City (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC20/306/R
Record Dates: First submitted 2020-07-09; First posted 2020-07-20 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; Acute Hypoxemic Respiratory Failure
Keywords: helmet nonivasive ventilation
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helmet group (Experimental): Patients will be allocated to helmet non-invasive ventilation
  Interventions: Device: Helmet non-invasive ventilation
- Control group (No Intervention): Patients will be allocated to standard of care

INTERVENTIONS:
Device: Helmet non-invasive ventilation — Patients will be allocated to helmet non-invasive ventilation
  Arms: Helmet group

SUMMARY:
Study hypothesis: Non-invasive positive pressure ventilation delivered by helmet will reduce 28-day all-cause mortality in patients with suspected or confirmed severe COVID-19 pneumonia and acute hypoxemic respiratory failure

DETAILED DESCRIPTION:
This will be a pragmatic parallel randomized control trial that will compare helmet nonivasive ventilation with standard of care to standard of care alone in 1:1 ratio. The trial will be implemented in multiple centers.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed COVID-19
* Aged ≥14 years old at the participating ICU. ICUs that use other age cut-off for adult patients will adhere to their local standard (16 or 18 years)
* Acute hypoxemic respiratory failure based on PaO2/FiO2 ratio <200 despite supplemental oxygen with a partial or non-rebreathing mask at a flow rate >10 L/min or above
* Intact airway protective gag reflex
* Able to follow instructions (e.g. squeeze hand on command, eye contact with care provider, stick out tongue on command, etc.)

Exclusion Criteria:

* Prior intubation during this hospital admission
* Cardiopulmonary arrest
* Glasgow coma scale <12
* Tracheostomy
* Upper airway obstruction
* Active epistaxis
* Requirement for more than one vasopressor to maintain mean arterial pressure > 65 mm Hg
* Pregnancy
* Imminent intubation
* Patients with do not intubate orders or equivalent
* Enrolled in another trial for which co-enrolment is not approved including trials on mechanical ventilation
* Patients already treated with helmet
* Patients with chronic carbon dioxide retention (PaCO2 >45)
* Previous enrolment in this trial
* The primary cause of respiratory failure is not heart failure as judged by the treating team

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28 days from randomization
  all cause mortality

SECONDARY OUTCOMES:
Intubation rate within 28 days | 28 days from randomization
  endotracheal intubation
ICU mortality | 180 days from randomization
  ICU death
Hospital mortality (censored at day 180) | 180 days from randomization
  hospital death
Hospital length of stay | 180 days from randomization
  length of stay in the hospital
ICU free days at day 28 | 28 days from randomization
  days not in ICU
Invasive ventilation-free days at day 28 | 28 days from randomization
  days without ventilator support
Renal replacement therapy-free days at day 28 | 28 days from randomization
  days without renal replacement therapy received
Vasopressor-free days at day 28 | 28 days from randomization
  days without vasopressor support
Safety outcome: skin pressure ulcers | 28 days from randomization
  presence of pressure ulcers
Safety outcome: barotrauma | 28 days from randomization
  incidence of barotrauma
Serious adverse events (including cardiovascular events and device complications) | 28 days from randomization
  reporting of abovementioned adverse events
180-day all-cause mortality | 180 days from randomization
  all cause mortality
Follow-up study: 180-day 5-level EQ-5D version | 180 days from randomization
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Yaseen Arabi, MD, Principal Investigator — King Abdulaziz Medical City - Riyadh
Locations (1):
- Intensive Care Department, King Abdulaziz Medical City, National Guard Health Affairs, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arabi YM, Al-Dorzi HM, Aldekhyl S, Al Qahtani S, Abdukahil SA, Al Qasim E, Al Harbi MK, Kharaba A, Albrahim T, Alshahrani MS, Al-Fares AA, Al Bshabshe A, Mady A, Al Duhailib Z, Algethamy H, Jose J, Al Mutairi M, Al Zumai O, Al Haji H, Alaqeily A, Al Wehaibi W, Al Aseri Z, Al-Omari A, Tlayjeh H, Al-Dawood A; Saudi Critical Care Trials Group. Long-term outcomes of patients with COVID-19 treated with helmet noninvasive ventilation or usual respiratory support: follow-up study of the Helmet-COVID randomized clinical trial. Intensive Care Med. 2023 Mar;49(3):302-312. doi: 10.1007/s00134-023-06981-5. Epub 2023 Feb 23. PMID 36820878
- [Derived] Arabi YM, Aldekhyl S, Al Qahtani S, Al-Dorzi HM, Abdukahil SA, Al Harbi MK, Al Qasim E, Kharaba A, Albrahim T, Alshahrani MS, Al-Fares AA, Al Bshabshe A, Mady A, Al Duhailib Z, Algethamy H, Jose J, Al Mutairi M, Al Zumai O, Al Haji H, Alaqeily A, Al Aseri Z, Al-Omari A, Al-Dawood A, Tlayjeh H; Saudi Critical Care Trials Group. Effect of Helmet Noninvasive Ventilation vs Usual Respiratory Support on Mortality Among Patients With Acute Hypoxemic Respiratory Failure Due to COVID-19: The HELMET-COVID Randomized Clinical Trial. JAMA. 2022 Sep 20;328(11):1063-1072. doi: 10.1001/jama.2022.15599. PMID 36125473
- [Derived] Arabi Y, Aldekhyl S, Al Qahtani S, Al-Dorzi HM, Abdukahil SA, Jose J, Al Harbi MK, Al Haji H, Al Mutairi M, Al Zumai O, Al Qasim E, Al Wehaibi W, Alshahrani M, Albrahim T, Mady A, Al Bshabshe A, Al Aseri Z, Al Duhailib Z, Kharaba A, Alqahtani R, Algethamy H, Alfaris O, Alnafel O, Al-Fares AA, Tlayjeh H. Helmet noninvasive ventilation for COVID-19 patients (Helmet-COVID): statistical analysis plan for a randomized controlled trial. Trials. 2022 Feb 2;23(1):105. doi: 10.1186/s13063-021-05988-x. PMID 35109898
- [Derived] Arabi YM, Tlayjeh H, Aldekhyl S, Al-Dorzi HM, Abdukahil SA, Al Harbi MK, Al Haji H, Al Mutairi M, Al Zumai O, Al Qasim E, Al Wehaibi W, Al Qahtani S, Al-Hameed F, Chalabi J, Alshahrani M, Albrahim T, Alharthy A, Mady A, Bin Eshaq A, Al Bshabshe AA, Al Aseri Z, Al Duhailib Z, Kharaba A, Alqahtani R, Al Ghamdi A, Altalag A, Alghamdi K, Almaani M, Algethamy H, Al Aqeily A, Al Baseet F, Al Samannoudi H, Al Obaidi M, Ismaiel YT, Al-Fares AA. Helmet Non-Invasive Ventilation for COVID-19 Patients (Helmet-COVID): study protocol for a multicentre randomised controlled trial. BMJ Open. 2021 Aug 26;11(8):e052169. doi: 10.1136/bmjopen-2021-052169. PMID 34446500